CLINICAL TRIAL: NCT01621412
Title: HIV Disclosure and Medication Adherence, a Pilot Study
Acronym: RSAD-VIH-11
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Swiss HIV Cohort Study (Network)
Responsible Party: Principal Investigator, Marie Schneider, Pharmacist, PhD, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Other Study IDs: RSAD-VIH-2011
Record Dates: First submitted 2012-05-31; First posted 2012-06-18 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infection
Keywords: Medication Adherence; HIV infection; Disclosure
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators believe that disclosure of HIV status could influence medication adherence. If disclosure leads to social support, adherence could be improved. This study purpose is to assess correlation between disclosure and medication adherence, and to describe people whose HIV status has been disclosed to.

DETAILED DESCRIPTION:
Pharmacists administer a questionnaire to each consecutive subject taking part in the adherence-enhancing program at the pharmacy of the Department of Ambulatory Care And Community Medicine in Lausanne. This questionnaire assesses disclosure, response to disclosure, and living situation.

Adherence is measured by electronic monitoring and pill count.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection
* Enrolled in the adherence-enhancing program

Exclusion Criteria:

* Inclusion visit
* Not french or english speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the adherence-enhancing program at ther pharmacy of Department of Ambulatory Care and Community Medicine in Lausanne
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Patient Adherence | 30 days before survey
  Electronic monitoring of adherence during 30 days before survey

SECONDARY OUTCOMES:
Patient Adherence | 90 days before survey
  Electronic monitoring of adherence during 90 days before survey

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule Schneider, PhD, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Aurélie Gertsch, PhD-Student, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Olivier Bugnon, Professor, Study Chair — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Matthias Cavassini, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Policlinique Médicale Universitaire, Lausanne, Canton of Vaud, Switzerland